CLINICAL TRIAL: NCT03897166
Title: Study of Volumetric, Radiomic and Anthropometric Characteristics in Trimodal Imaging (Positron Emission Tomography, Computed Tomography, Magnetic Resonance Imaging) Before Radiotherapy
Brief Title: Trimodal Imaging Before Radiotherapy
Acronym: TRIMODAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHB 17.02
Record Dates: First submitted 2019-02-05; First posted 2019-04-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trimodality Imaging (Experimental): Positron Emission Tomography coupled with Computed Tomography computed coupled with Magnetic Resonance Imaging and whole-body Biphoton Absorptiometry
  Interventions: Device: Trimodality

INTERVENTIONS:
Device: Trimodality — Positron Emission Tomography coupled with Computed tomography and immediately followed by Magnetic Resonance Imaging

SUMMARY:
In oncology, personalized medicine is progressing by providing increasingly tumor- and patient-specific care. Thus, medical imaging allows precise morphological and functional characterization of the tumor by volume measurements, used in particular in radiotherapy to define the macroscopic tumor volume (GTV), and radiomic measurements that correspond to a recent concept of extraction of textural parameters and/or tumor shape (tumor heterogeneity, tumor invasiveness...). Precise characterization of the patient is also possible by anthropometric measurements (measurements of total muscle mass, visceral adipose tissue mass...) which can be important predictive and prognostic factors and which are generally estimated more accurately in imaging than by using mathematical formulas.

However, these measurements are partly dependent on the imaging acquisition mode (PET, CT or MRI). The volume measurements, and therefore the GTV, are thus different depending on the imaging used. Studying these differences is important because no single imaging technique encompasses all potential GTV regions but, on the other hand, a combination of anatomical and functional information could improve tumor delineation. Beyond this volume analysis, the extraction of radiomic characteristics seems very promising in radiotherapy with however many limitations to be overcome, linked in particular to the data acquisition mode. Concerning anthropometric measurements, CT and MRI have become essential techniques for precise anatomical quantification, particularly of lean mass, visceral adipose tissue or muscle mass, but automatic measurement techniques for these parameters have yet to be defined, particularly during CT or MRI acquisitions associated with PET for attenuation correction.

To identify useful volume, radiomic and anthropometric characteristics, medical imaging thus requires prospective cohorts of patients with comparable cancer histologies and standardized images acquired by different modalities (e. g. PET, CT or MRI) during the pre-treatment assessment before similar treatments.

The purpose of this study is to create a prospective cohort to study volume, radiomic and anthropometric characteristics by taking advantage of the recent installation of MRI in the medical imaging department of the Henri Becquerel Cancer Center (HBCC), Rouen, France, allowing PET/MRI to be performed and by taking advantage of the collaboration between the radiotherapy and medical imaging departments of the HBCC.

DETAILED DESCRIPTION:
The purpose of this study is to create a prospective cohort to study volume, radiomic and anthropometric characteristics. For that 60 patients will be included before treatment by radiotherapy.

Patients will benefit from a detailed pre-therapeutic imaging assessment with trimodal acquisitions (CT/MRI/PET with 18F-FDG) before radiotherapy and in radiotherapeutic position according to the "CRAI" (for "Centre Régional de thérapie Assistée par l'Imagerie") acquisition protocol, innovative in trimodality.

This initial imaging assessment will be supplemented by a whole-body biphoton absorptiometry which will be used as a reference examination for certain anthropometric parameters. This examination will be carried out at the Rouen University Hospital in the Rheumatology Department

ELIGIBILITY:
Inclusion Criteria:

* Positron Emission Tomography before radiotherapy
* More than 18 years
* PS 0 to 1
* Signed Inform consent Form

Exclusion Criteria:

* Contraindication to Magnetic resonance Imaging
* More than 150 kgs
* Pregnancy or child bearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Difference of volumes estimated by geometric indices with the three techniques | 2 weeks
  The volumes studied will be defined for each imaging modality individually and in combination, taking into account several modalities at the same time

SECONDARY OUTCOMES:
Determination of methods to measure radiomics parameters | 2 weeks
  the comparison of the different parameters obtained with a study of intra-modality and inter-modality correlations with algorithm to compare trimodality with the reference techniques
quality of the MRI PET attenuation correction: differences in SUVmax, SUVpeak and SUVmean | 2 weeks
  the calculation of differences in SUVmax, SUVpeak and SUVmean

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Decazes, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No